CLINICAL TRIAL: NCT01845428
Title: Assessment of the Efficacy of Lipid-lowering Agents to Limit Lipid Oxidation and Activation of the Clotting System in Patients With the Nephrotic Syndrome: a Pilot Study.
Brief Title: Lipid Lowering Agents to Limit Lipid Oxidation and Activation of Clotting System in Nephrotic Syndrome
Acronym: OxLDL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12-0789; U54DK083912 (NIH)
Record Dates: First submitted 2013-04-24; First posted 2013-05-03 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Nephrotic Syndrome; Hyperlipidemia
Keywords: nephrotic; hyperlipidemia; oxLDL; kidney
MeSH Terms: conditions — Nephrotic Syndrome; Hyperlipidemias | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pravastatin (Other): All participants will receive pravastatin 20mg daily
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — After collecting baseline plasma samples, participants will receive pravastatin 20mg daily. After 6 weeks, we will collect samples and safety data. Subsequent statin therapy will be at the discretion of the treating physician.
  Other Names: Pravachol

SUMMARY:
The purpose of this research study is to learn if using statin in patients with nephrotic syndrome could lower the risk of blood clots. Nephrotic syndrome is a collection of signs and symptoms that occur when the glomeruli -the tiny filters that work in the kidney- leak protein in the urine.

One of the symptoms associated with nephrotic syndrome is hyperlipidemia: too much bad cholesterol (LDL). This bad cholesterol could be linked to the increased risk of blood clots in patients with nephrotic syndrome. The study doctors would like to see if taking a statin drug to reduce the amount of bad cholesterol could reduce the risk of blood clots.

DETAILED DESCRIPTION:
Venous thromboembolic (VTE) events are common in the nephrotic syndrome (NS) occurring in up to 30% of patients when systematically screened. The investigator proposes to explore a novel mechanism for the increased clot formation in NS. To date, the only consistently identified underlying risk factor for VTEs is severe hypoalbuminemia related to the NS. The underlying pathophysiology related to VTE in NS remains poorly understood and has previously been ascribed to dysregulation of pro- and anticoagulant clotting factors due to urinary protein losses and reflected by the low serum albumin. However, the direct evidence for this mechanism is inconsistent and relatively poor. Another feature of NS is that of severe hyperlipidemia which also correlates with hypoalbuminemia. In other severely hyperlipidemic states (e.g. Familial Hypercholesterolemia), the level of oxidized low-density lipoprotein (oxLDL) is markedly elevated. Forms of oxidized LDL interact with monocytes and macrophages leading to expression of Tissue Factor (TF), a procoagulant molecule. Furthermore, monocytes and macrophages activated in this fashion also release microparticles, small cell-membrane derived vesicles, that also express TF and participate in initiating intravascular clot formation. the investigator hypothesizes that the hyperlipidemia of the nephrotic syndrome leads to elevations in oxidized LDL and in turn, elevations in microparticle Tissue Factor (MP-TF) and its activity. The investigator also hypothesizes that serum albumin levels will inversely correlate with hyperlipidemia as well as oxLDL levels and MP-TF activity. Here, the investigator will study the effect of treatment with HMGCoA reductase inhibitors (statins) on ox LDL and MP-TF activity patients with NS.

ELIGIBILITY:
Inclusion Criteria:• Prevalent or incident patients of either sex, ages 18-70, with Membranous Nephropathy (MN) , Focal Segmental GlomeruloSclerosis (FSGS), or Minimal Change Disease (MCD).

* Proteinuria ≥ 3.0 g/day by 24hr urine collection or urine protein/creatinine ratio ≥ 2.
* Hyperlipidemia as defined by fasting or direct LDL ≥ 150 mg/dl. -

Exclusion Criteria:Inability or unwillingness to comply with the study protocol and follow-up visits.

Patients unable to provide written consent will be excluded.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in Microparticle tissue factor (MP-TF) activity | tested at baseline and week 6
  The investigator will measure MP-TF activity . Microparticles will be isolated from platelet-free plasma (PFP) in a two-step sequential ultracentrifugation (20,000xg) process. Following the addition of Factor VIIa, Factor X and CaCl2, FXa generation is measured. Recombinant human relipidated TF will be used as a standard. TF-dependent plasma coagulation activity (PCA)generation is calculated by subtracting PCA generated in the presence of blocking antibodies from the amount of total PCA generated in the presence of an IgG control. The use of MP-TF activity as an outcome measure is unique in that it reflects both the pathophysiology and is a measure of PCA that correlates with VTE events

SECONDARY OUTCOMES:
Changes in plasma coagulation activation | baseline and week6
  the investigator will also perform other more routine measures of plasma coagulation activation to determine the overall effect of hyperlipidemia in NS that may include TF-independent mechanisms.
  Thrombin-antithrombin complexes (TAT) also provide information regarding the downstream effect of Tissue Factor in the coagulation cascade.
  1. D-Dimer measurement - human D-Dimer ELISA
  2. Thrombin-antithrombin complexes (TAT) -
  Other covariates:
  Fasting lipid profile (including direct LDL measurement), serum albumin, proteinuria (by urine protein/creatinine ratio), estimated Glomerular Filtration Rate (eGFR), immunosuppressive therapy, age, sex, race.

CONTACTS AND LOCATIONS:
Overall Officials: Vimal Derebail, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Unc Kidney Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: general web site of UNC Kidney Center — https://unckidneycenter.org/